CLINICAL TRIAL: NCT00701181
Title: A Phase II Prospective, Randomized, Multi-Center, Diabetic Macular Edema Dose Ranging, Comparator Study Evaluating The Efficacy And Safety Of PF-04523655 Versus Laser Therapy (DEGAS)
Brief Title: Study Evaluating Efficacy and Safety of PF-04523655 Versus Laser in Subjects With Diabetic Macular Edema
Acronym: DEGAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Quark Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B0451004
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Diabetic Retinopathy; Diabetes Complications
Keywords: Phase II; Prospective; Randomized; Diabetic Macular Edema; PF-04523655; Laser
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Complications | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Laser (Active Comparator): This is a procedure - not a drug intervention.
  Interventions: Procedure: Laser Treatment
- PF-04523655 (High) (Experimental)
  Interventions: Drug: PF-04523655 high
- PF-04523655 middle (Experimental)
  Interventions: Drug: PF-04523655 middle
- PF-04523655 low (Experimental)
  Interventions: Drug: PF-04523655 low

INTERVENTIONS:
Procedure: Laser Treatment — Necessity of laser treatment is assessed every three months.
  Arms: Laser
Drug: PF-04523655 high — 3 mg intravitreal injection
  Arms: PF-04523655 (High)
Drug: PF-04523655 middle — 1 mg intravitreal injection
  Arms: PF-04523655 middle
Drug: PF-04523655 low — 0.4 mg intravitreal injection
  Arms: PF-04523655 low

SUMMARY:
To evaluate the effectiveness of study drug in improving visual acuity compared to laser treatment in the patients with diabetic macular edema

DETAILED DESCRIPTION:
DEGAS termination decision date was December 17, 2010. Rationale: the objectives of the study could no longer be achieved. The study was not terminated for safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus (Type 1 or Type 2) Showing Diabetic Macular Edema in the Eye.

Exclusion Criteria:

* Proliferative Diabetic Retinopathy in the Study Eye.
* Subjects Receiving Concomitant Intravitreal Anti-VEGF Therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in the Best Corrected Visual Acuity Score | Month 24

SECONDARY OUTCOMES:
Mean Changes in NEI-VFQ-25 Composite Score from Baseline | Month 24, 36
Plasma Concentration of PF-04523655 | Week 1
Percent of Subjects Gaining Letters in the Best Corrected Visual Acuity Score from Baseline. | Month 24, 36
Incidence and Severity of Ocular and Systemic Adverse Events, as Identified by Ophthalmic Examination | Month 24, 36
Mean Change from Baseline in the Best Corrected Visual Acuity Score | Month 36
Mean Changes in Area of Fluorescein Leakage from Baseline | Month 24, 36
Percent of Subjects Losing Letters in the Best Corrected Visual Acuity Score from Baseline. | Month 24, 36
Mean Changes in Retinal Thickness from Baseline | Month 24, 36
Mean Changes in Macular Volume from Baseline | Month 24, 36

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (23):
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Meza, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Mountain View, California
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, ‘Aiea, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Portsmouth, New Hampshire
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, High Point, North Carolina
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Rapid City, South Dakota
  - Pfizer Investigational Site, Corpus Christi, Texas
- Pfizer Investigational Site, Glostrup Municipality, Denmark
- Germany (3):
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Münster
- India (4):
  - Pfizer Investigational Site, Bhubaneshwar, Odisha
  - Pfizer Investigational Site, Ahmedabad
  - Pfizer Investigational Site, Bangalore
  - Pfizer Investigational Site, New Delhi
- Israel (5):
  - Pfizer Investigational Site, Kfar Saba
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
  - Pfizer Investigational Site, Ẕerifin
- Italy (4):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Udine
- Pfizer Investigational Site, Lima, Lima Province, Peru
- United Kingdom (5):
  - Pfizer Investigational Site, Frimley, Camberley, Surrey
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Southampton

REFERENCES:
- [Derived] Nguyen QD, Schachar RA, Nduaka CI, Sperling M, Basile AS, Klamerus KJ, Chi-Burris K, Yan E, Paggiarino DA, Rosenblatt I, Aitchison R, Erlich SS; DEGAS Clinical Study Group. Dose-ranging evaluation of intravitreal siRNA PF-04523655 for diabetic macular edema (the DEGAS study). Invest Ophthalmol Vis Sci. 2012 Nov 15;53(12):7666-74. doi: 10.1167/iovs.12-9961. PMID 23074206
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0451004&StudyName=Prospective%2C%20Randomized%2C%20Multi-Center%2C%20Comparator%20Study%20Evaluating%20Efficacy%20and%20Safety%20of%20PF-04523655%20versus%20Laser%20in%20Subjects%20with%20Diab